CLINICAL TRIAL: NCT05064332
Title: A PHASE 1, OPEN LABEL, FIXED SEQUENCE STUDY TO ESTIMATE THE EFFECT OF MULTIPLE DOSE PF-06650833 ON THE PHARMACOKINETICS OF SINGLE DOSE ORAL CONTRACEPTIVE STEROIDS IN HEALTHY FEMALE PARTICIPANTS
Brief Title: A Study To Estimate The Effect of PF-06650833 On The Pharmacokinetics (PK) of Oral Contraceptive (OC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: B7921026
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Results first posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2022-11

CONDITIONS: Healthy
MeSH Terms: interventions — 1-(((2S,3S,4S)-3-ethyl-4-fluoro-5-oxopyrrolidin-2-yl)methoxy)-7-methoxyisoquinoline-6-carboxamide; Ethinyl Estradiol; Contraceptives, Oral

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OC only (Experimental): Subjects will receive a single dose of an oral contraceptive during the first period of the study
  Interventions: Drug: Ethinyl estradiol (EE) and levonogestrel (LN)
- PF-06650833 + OC (Experimental): Subjects will receive PF-06650833 every day for 11 days and a single dose of an oral contraceptive on day 10.
  Interventions: Drug: PF-06650833; Drug: Ethinyl estradiol (EE) and levonogestrel (LN)

INTERVENTIONS:
Drug: PF-06650833 — 400 mg by mouth (PO) Once daily (QD) for 11 days
  Arms: PF-06650833 + OC
Drug: Ethinyl estradiol (EE) and levonogestrel (LN) — Single dose of Oral tablet containing 30 ug EE and 150 ug of LN
  Other Names: Oral contraceptive (OC)

SUMMARY:
This is a Phase 1, open label, fixed sequence study of the effect of multiple dose PF-06650833 on single dose OC PK in healthy female subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment in the study:

1. Healthy female subjects
2. Female subjects of non childbearing potential must meet at least 1 of the following criteria:

   1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state;
   2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   3. Have medically confirmed ovarian failure.

   All other female subjects (including female subjects with tubal ligations) are considered to be of childbearing potential and will be eligible with adequate contraceptive usage.
3. Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
3. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
4. Any current evidence of untreated active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB).
5. History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing
6. Benign ethnic (cyclic) neutropenia.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Qps-Mra, Llc, South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7921026

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened 28 days prior to the first dose of study intervention in Period 1 and reported to the clinical research unit the day prior to Day 1 dosing in Period 1.
Pre-assignment Details: The study consisted of 2 periods in a single fixed sequence. Period 1 was immediately followed by Period 2 with no washout. A total of 10 participants were enrolled in the study.
Groups:
- Oral Contraceptive (OC) Then PF-06650833+ OC: Participants received a single oral dose of OC, containing ethinyl estradiol (EE) 30 microgram (mcg) and levonorgestrel (LN) 150 mcg on Day 1 Period 1. After completion of Period 1, participants orally received PF-06650833 400 milligram (mg) once daily (QD) on Days 1-11 of Period 2 and a single oral dose of OC, containing EE 30 mcg and LN 150 mcg on Day 10 Period 2.
Period: Period 1
Arm/Group | Oral Contraceptive (OC) Then PF-06650833+ OC
Started | 10
Completed | 10
Not Completed | 0
Period: Period 2
Arm/Group | Oral Contraceptive (OC) Then PF-06650833+ OC
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population defined as all participants enrolled to study intervention and who took at least 1 dose of study intervention.
Groups:
- OC Then PF-06650833+ OC: Participants received a single oral dose of OC, containing EE 30 mcg and LN 150 mcg on Day 1 Period 1. After completion of Period 1, participants orally received PF-06650833 400 mg QD on Days 1-11 of Period 2 and a single oral dose of OC, containing of EE 30 mcg and LN 150 mcg on Day 10 Period 2.
Arm/Group | OC Then PF-06650833+ OC
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) for Ethinyl Estradiol
Description: AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration. AUClast for EE was determined using linear/Log trapezoidal method.
Time Frame: Predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36 and 48 hours post OC dose in Periods 1 and 2
Population: The PK parameter analysis population was defined as all participants that received at least 1 dose of study intervention and had at least 1 of the PK parameters of primary interest reported in at least 1 period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour per milliliter (pg*hr/mL)
Groups:
- Period 1: Oral Contraceptive: Participants received a single oral dose of OC, containing EE 30 mcg and LN 150 mcg on Day 1 Period 1.
- Period 2: PF-06650833 + Oral Contraceptive: Participants orally received PF-06650833 400 mg QD on Days 1-11 of Period 2 and a single oral dose of OC, containing of EE 30 mcg and LN 150 mcg on Day 10 Period 2.
Arm/Group | Period 1: Oral Contraceptive | Period 2: PF-06650833 + Oral Contraceptive
Number analyzed (Participants) | 10 | 10
picogram*hour per milliliter (pg*hr/mL) | 812.3 (25) | 823.9 (26)
Statistical Analysis 1: Comparison: Period 1: Oral Contraceptive vs Period 2: PF-06650833 + Oral Contraceptive; OC alone as the Reference and co-administration of PF-06650833 and OC as the Test. Natural log transformed AUClast was analyzed using a mixed effects model with treatment as a fixed effect and participant as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence intervals (CIs) were obtained from the model and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Other; Ratio of Adjusted Geometric Means = 101.43, 90% CI 2-sided [93.01 to 110.61]

2. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration for Levonorgestrel
Description: AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration. AUClast for LN was determined using linear/Log trapezoidal method.
Time Frame: Predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36 and 48 hours post OC dose in Periods 1 and 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hr/mL
Arm/Group | Period 1: Oral Contraceptive | Period 2: PF-06650833 + Oral Contraceptive
Number analyzed (Participants) | 10 | 10
pg*hr/mL | 31510 (39) | 34190 (41)
Statistical Analysis 1: Comparison: Period 1: Oral Contraceptive vs Period 2: PF-06650833 + Oral Contraceptive; OC alone as the Reference and co-administration of PF-06650833 and OC as the Test. Natural log transformed AUClast was analyzed using a mixed effects model with treatment as a fixed effect and participant as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Other; Ratio of Adjusted Geometric Means = 108.51, 90% CI 2-sided [98.85 to 119.11]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) for Ethinyl Estradiol
Description: Cmax was defined as maximum plasma concentration. Cmax for EE was observed directly from data.
Time Frame: Predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36 and 48 hours post OC dose in Periods 1 and 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram per milliliter (pg/mL)
Arm/Group | Period 1: Oral Contraceptive | Period 2: PF-06650833 + Oral Contraceptive
Number analyzed (Participants) | 10 | 10
picogram per milliliter (pg/mL) | 84.00 (38) | 79.86 (26)
Statistical Analysis 1: Comparison: Period 1: Oral Contraceptive vs Period 2: PF-06650833 + Oral Contraceptive; OC alone as the Reference and co-administration of PF-06650833 and OC as the Test. Natural log transformed Cmax was analyzed using a mixed effects model with treatment as a fixed effect and participant as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence intervals (CIs) were obtained from the model and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Other; Ratio of Adjusted Geometric Means = 95.07, 90% CI 2-sided [84.44 to 107.04]

4. Primary Outcome: Maximum Plasma Concentration for Levonorgestrel
Description: Cmas was defined as maximum plasma concentration. Cmax for LN was observed directly from data.
Time Frame: Predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36 and 48 hours post OC dose in Periods 1 and 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Period 1: Oral Contraceptive | Period 2: PF-06650833 + Oral Contraceptive
Number analyzed (Participants) | 10 | 10
pg/mL | 3468 (56) | 4092 (53)
Statistical Analysis 1: Comparison: Period 1: Oral Contraceptive vs Period 2: PF-06650833 + Oral Contraceptive; OC alone as the Reference and co-administration of PF-06650833 and OC as the Test. Natural log transformed Cmax was analyzed using a mixed effects model with treatment as a fixed effect and participant as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Other; Ratio of Adjusted Geometric Means = 117.99, 90% CI 2-sided [101.82 to 136.73]

5. Secondary Outcome: Number of Participants With Treatment Emergent Treatment-Related Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An serious adverse event (SAE) was defined as an AE: 1. resulting in death, 2. was life-threatening, 3. required inpatient hospitalization or prolongation of existing hospitalization, 4. resulted in persistent disability, 5. was a congenital anomaly/birth defect, or considered to be an important medical event. Treatment-related AE was any untoward medical occurrence attributed to study intervention in a participant who received study intervention. Treatment-emergent are events between first dose of study intervention and up to 35 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the first dose up to 35 days after the last dose of study intervention
Population: The safety analysis set was defined as all participants enrolled to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Period 2: PF-06650833: Participants orally received PF-06650833 400 mg QD on Days 1-10 of Period 2.
- Period 2: PF-06650833 + Oral Contraceptive: Participants received a single oral dose of OC, containing of EE 30 mcg and LN 150 mcg on Day 10 Period 2 and a single oral dose of PF-06650833 400 mg on Day 11 Period 2.
Arm/Group | Period 1: Oral Contraceptive | Period 2: PF-06650833 | Period 2: PF-06650833 + Oral Contraceptive
Number analyzed (Participants) | 10 | 10 | 10
Participants
  Treatment-related AEs | 0 | 0 | 0
  Treatment-related SAEs | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events by Severity
Description: An AE was any untoward medical occurrence attributed to study intervention in a participant who received study intervention. AEs are classified according to the severity in 3 categories. a) mild - AEs does not interfere with participant's usual function; b) moderate - AEs interferes to some extent with participant's usual function; c) severe - AEs interferes significantly with participant's usual function. Only those categories in which at least 1 participant had data were reported.
Time Frame: From the first dose up to 35 days after the last dose of study intervention
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Oral Contraceptive | Period 2: PF-06650833 | Period 2: PF-06650833 + Oral Contraceptive
Number analyzed (Participants) | 10 | 10 | 10
Participants
  Nausea (mild) | 0 | 1 | 0
  Toothache (mild) | 0 | 0 | 1
  Headache (mild) | 0 | 1 | 0
  Pruritus (mild) | 0 | 2 | 0

7. Secondary Outcome: Number of Participants With Categorical Vital Signs Data of Potential Clinical Concern
Description: Systolic blood pressure (BP), diastolic BP and supine pulse rate measurements meeting the criteria of potential clinical concern were summarized by treatment using categories as defined: Systolic BP min. <90 mmHg; Systolic BP max. decrease ≥30 or max. increase ≥30; Diastolic BP min. <50 mmHg; Diastolic BP max. decrease ≥20 or max. increase ≥20; Supine pulse rate min. <40 bpm or max. >120 bpm.
Time Frame: Day 1 for Period 1 and Day 1, Day 10, Day 12 for Period 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Oral Contraceptive | Period 2: PF-06650833 + Oral Contraceptive
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities of Potential Clinical Concern
Description: Hematology (hemoglobin, hematocrit, erythrocytes [Ery.], Ery.mean corpuscular volume, Ery.mean corpuscular hemoglobin, platelets, leukocytes, lymphocytes, neutrophils, basophils, eosinophils, monocytes); clinical chemistry (bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, protein, albumin, urea nitrogen, creatinine, urate, sodium, potassium, chloride, calcium, bicarbonate, glucose, creatine kinase); and urinalysis (pH, glucose, ketones, protein, hemoglobin, urobilinogen, bilirubin, nitrite, leukocyte esterase, Ery., leukocytes, epithelial cells, casts and bacteria) tests were assessed. Only those categories, in which at least 1 participant had data were reported.
Time Frame: Day 10, Day 12 for Period 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Period 2: PF-06650833 + Oral Contraceptive
Number analyzed (Participants) | 10
Participants
  Urine Hemoglobin ≥1 | 5
  Leukocyte Esterase ≥1 | 2

ADVERSE EVENTS:
Time Frame: From the first dose up to 35 days after the last dose of study intervention.
Description: MedDRA 24.1 coding dictionary was applied for all AE tables. The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Period 1: Oral Contraceptive | Period 2: PF-06650833 | Period 2: PF-06650833 + Oral Contraceptive
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 2/10 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Oral Contraceptive (N=10) | Period 2: PF-06650833 (N=10) | Period 2: PF-06650833 + Oral Contraceptive (N=10)
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT05064332/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT05064332/SAP_001.pdf